CLINICAL TRIAL: NCT01049087
Title: Comparison of Plasma Volume Determination by 99mTc-labeled Albumin and 125I-labeled Albumin
Brief Title: Plasma Volume Determination by 99mTc-labeled Albumin and 125I-labeled Albumin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Peter Kramshoj Bonfils, University Hospital Koge, Department of Clinical Physiology and Nuclear Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: SJ-112
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: plasma volume; technetium-labeled albumin; radioiodine-labeled albumin; Healthy volunteers
MeSH Terms: interventions — Plasma Volume

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Plasma volume determination (99mTc-albumin) — The test is performed using 5MBq technetium-labeled albumin (99mTc-albumin-Vasculosis) with several postinjection samples for accurate zero-time extrapolation.
Radiation: Plasma volume determination (125I-albumin) — The test is performed using 0.2MBq 125iodine-labeled albumin (125I-albumin) with several postinjection samples for accurate zero-time extrapolation.

SUMMARY:
The purpose of the present study is to compare plasma volume determination by 99mTc-labeled albumin with 125I-labeled albumin. Fifteen subjects will be enrolled. The hypothesis is that plasma volume determined by the different methods are the same.

DETAILED DESCRIPTION:
For many years, radioiodinated albumin has been "the golden standard" for measurement of plasma volume. There are a number of clinical situations in which a nuclide with a shorter half-life would be preferred. Furthermore, due to periodic lapses in the availability in the delivery of 125I-labeled albumin, there is a need to evaluate another nuclide as a tracer for plasma volume determination.

99mTc-labeled albumin is easily prepared by a simple and reproducible method with a high labeling efficiency and short half-life.

In this study, we want to compare plasma volume determined by 99mTc-labeled albumin with plasma volume determined by 125I-albumin (golden standard). In both procedures, plasma volume is estimated from multiple postinjection samples for accurate zero-time extrapolation in order to correct for leakage of labeled albumin from the vascular compartment.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 27 kg/m2
* Written informed consent

Exclusion Criteria:

* Hypertension (140/90 mmHg)
* Diabetes mellitus
* Any use of medication
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Plasma volume determined by 99mTc-labeled albumin and 125I-labeled albumin | January 2011

SECONDARY OUTCOMES:
Rates of loss of 99mTc-labeled albumin and 125I-labeled albumin from the circulation | January 2011

CONTACTS AND LOCATIONS:
Overall Officials: Steen Levin, MD, DMSc, Study Chair — Zealand University Hospital; Peter K Bonfils, MD, Principal Investigator — Zealand University Hospital; Knud H Stokholm, MD, Study Director — Zealand University Hospital
Locations (1):
- University Hospital Koge, Department of Clinical Physiology and Nuclear Medicine, Køge, Denmark